CLINICAL TRIAL: NCT04896333
Title: Acceptability in Dialogues Between the Robot EBO and Older Adults
Brief Title: Acceptability in Dialogues With the Robot EBO
Status: Completed | Type: Observational
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Elisa María Garrido Ardila, Clinical Professor, University of Extremadura
Other Study IDs: 128/2018
Record Dates: First submitted 2021-05-02; First posted 2021-05-21 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Nervous System Diseases
Keywords: Nervous System Diseases; acceptability; Robot
MeSH Terms: conditions — Nervous System Diseases | interventions — Drug Interactions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robot interaction: EBO is a robotic platform consisting of the following: A screen display capable of generating emotions (sadness, joy, neutral, anger, disgust and surprise), RGB camera, basic navigation system.
  EBO must be controlled by a teleoperator through a user-friendly and simple interface. Communication should be as immediate as possible, as well as predefined. In any case, the dialogue flow can be modified if necessary. The interface, at the same time, allows the possibility of sending emotions and small movements to the robot, to accompany the dialogue with certain elements of emotionality.
  The experiment replicates the Wizard of Oz technique. In this technique, the human tele-operator controls the robot without the person noticing it as he is in another room. For this purpose, a user interface will be displayed on the teleoperator's terminal and the commands will be reproduced by the EBO robot
  Interventions: Other: Interaction and exposure with the Robot EBO

INTERVENTIONS:
Other: Interaction and exposure with the Robot EBO — The participants will interact with the Robot EBO. The robot will be control by an operator that will conduct a dialogue. The dialogue will include questions related to the social, leisure, activities of daily living and informative areas.

SUMMARY:
This is a descriptive observational study (first results cross-sectional study, second results longitudinal study). The participants of the study will be exposed to a dialogue with the robot EBO. The user and the therapist's acceptability of the robot, the robot-user interaction during the conversation and the conversation parameters will be assessed.

DETAILED DESCRIPTION:
This is a descriptive observational study (first results cross-sectional study, second results longitudinal study). The participants of the study will be exposed to a dialogue with the robot EBO. The user and the therapist's acceptability of the robot will be measure. Also the robot-user interaction during the conversation and the conversation parameters will be assessed. The assessements will be done at week 0 and at week 3. During weeks 1 and 2 the robot will be present in the therapeutic activities of the center.

ELIGIBILITY:
Inclusion Criteria:

* Users of socio-health centers in Extremadura (Spain).
* Patients with neurological pathology diagnosed by a specialist doctor.
* Over 65 years of age
* Minimental State Examination with a score greater than or equal to 21 (mild-moderate cognitive impairment).

Exclusion Criteria:

* Severe cognitive impairment
* Language impairment that prevents the use of verbal communication.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population of study will be patients with neurological disorders who receive rehabilitation treatment in socio-health centers in Extremadura (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Robot-user interaction during the conversation: Conversation topic that most motivates the user or with which the user most interacts with the robot measured by recording and viewing the conversation | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Robot-user interaction during the conversation measured by recording and viewing the conversation
Robot-user interaction during the conversation: attempts to touch the robot by the patient measured by recording and viewing the conversation | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Robot-user interaction during the conversation measured by recording and viewing the conversation
Robot-user interaction during the conversation: times the user asks the robot questions measured by recording and viewing the conversation | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Robot-user interaction during the conversation measured by recording and viewing the conversation.
Robot-user interaction during the conversation: emotions that the conversation provokes in the patient measured by recording and viewing the conversation | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Robot-user interaction during the conversation measured by recording and viewing the conversation: emotions that the conversation provokes in the user (Standard, happy, sad, angry)
Robot-user interaction during the conversation: number of total interactions measured by recording and viewing the conversation | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Robot-user interaction during the conversation measured by recording and viewing the conversation.
Conversation parameters: time of the dialogue measured by the robot's register | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Conversation parameters measured by the robot's register
Conversation parameters: speed of response measured by the robot's register | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Conversation parameters (measured by the robot's register): speed of response (time taken by the patient to respond)
Conversation parameters: eye contact and patient's attention measured by the robot's register | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Conversation parameters (measured by the robot's register): eye contact with the robot and the attention of the patient to follow the conversation.
Conversation parameters: repetition of questions measured by the robot's register | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  Conversation parameters (measured by the robot's register): number of times the patient needed to be asked a question again.
User acceptability of the robot with the Technology Acceptance Model questionnaire | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  User acceptability of the robot measured with the Technology Acceptance Model. This scale has good validity and reliability, with a Cronbach's alpha value above 0.8 (Alenazy, Mugahed Al-Rahmi, & Khan, 2019). It assesses the following dimensions relating to the technology product:
  * Perceived ease of use: the extent to which users believe that using a particular system would improve their performance.
  * Perceived usefulness: the extent to which the individual believes that using the system will be effortless
  * Attitude towards use
  * Relevance
  A higher scores indicates a higher acceptability.
User acceptability of the robot measures with an specific designed questionnaire | Measured at the exposure/dialogue of the patient with the robot EBO during the intervention
  User acceptability of the robot measured with a questionnaire designed by the authors of the study. The questionnaire has 10 items that evaluate the acceptability of the robot by the user. This 10 questions have 3 choice answer with the options being yes, no, I don not know. There is one open question to collect qualitative data a¡regarding the dialogue and the acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Cáceres, Spain